CLINICAL TRIAL: NCT04900246
Title: Evaluation of Different Methods for the Diagnosis of Primary Caries Lesions: Study Protocol for a Randomized Controlled Clinical Trial
Brief Title: Evaluation of Different Methods for the Diagnosis of Primary Caries Lesions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: iTero
Record Dates: First submitted 2021-05-11; First posted 2021-05-25 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Caries Class II
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Visual Inspection + BWX Radiographic Assessment + Assessment of the iTero Element 5D scan (Experimental): In this group, the evaluations will follow this order. First the visual inspection, then the bitewing X-ray assessment and, lastly, the iTero assessment.
  Interventions: Procedure: Visual Inspection; Radiation: BWX Radiographic Assessment; Device: Assessment of the iTero Element 5D scan
- Visual Inspection + Assessment of the iTero Element 5D scan + BWX Radiographic Evaluation (Experimental): In this group, the evaluations will follow this order. First the visual inspection, then the iTero assessment and, lastly, the bitewing X-ray assessment.
  Interventions: Procedure: Visual Inspection; Radiation: BWX Radiographic Assessment; Device: Assessment of the iTero Element 5D scan

INTERVENTIONS:
Procedure: Visual Inspection — The examiners will evaluate the surfaces included in the study independently and without knowledge of the results of the other examiner, after prophylaxis, using a mouth mirror and a WHO probe or "Ball point". The evaluations will be carried out in a dental chair with the aid of a reflector. The teeth will be examined moist, and afterwards, they will be dried for 5 seconds with the use of a triple syringe.
  For visual inspection, the International Caries Detection and Assessment System (ICDAS) evaluation system will be used. Complete ICDAS has seven categories, the first for healthy teeth (code 0) and the next two for limited enamel caries, white/brown stain (codes 1 and 2). The following two categories (codes 3 and 4) are considered to be caries that extend to the enamel without exposed dentin. And the two remaining categories (codes 5 and 6), are considered caries with exposed dentin.
Radiation: BWX Radiographic Assessment — Participants will be radiographed with a digital X-ray device (DIOX-602, Micro Imagem, Indaiatuba, Brazil) with a regulation of 60 kV and 2 mA and exposure time of 0.10s. The technique used will be the interproximal/bitewing (BWX), with the FIT T1 Digital Sensor (external dimensions: 36.7mm x 24.3mm/sensitive area dimensions: 30.0mm x 20.0mm - 600mm²) and the sockets will be standardized with use of Han-Shin radiographic positioners (Jon, São Paulo, Brazil).
Device: Assessment of the iTero Element 5D scan — For scanning, the iTero 5D (Align Technology) equipment featuring NIRI Technology will be used. The Infrared Imaging Technology (NIRI) is a diagnostic tool that allows the detection of interproximal and occlusal caries in several stages, from the initial enamel caries to lesions in the amelo-dentin junction, without the use of ionizing radiation. Infrared is the region of the electromagnetic spectrum between 0.7 and 2.0 micrometers (µm). The iTero Element 5D imaging system uses wavelength light (= 850 nm) in an electromagnetic spectrum that, in interaction with the hard tooth tissue, provides additional data on its structure.

SUMMARY:
According to the World Health Organization (WHO), dental caries is considered one of the major pediatric health problems worldwide, due to its high prevalence and incidence. Therefore, the early diagnosis of caries lesions is a fundamental procedure for building the treatment plan, aiming at prevention, minimal intervention and the promotion of oral health. The present study aims to evaluate, through a randomized and controlled clinical study, which is the best strategy for diagnosing primary caries lesions located in the interproximal region in individuals aged from 4 to 10 years. Diagnostic methods will be analyzed and compared: visual clinical examination using the International Caries Detection and Assessment System (ICDAS), iTero Element 5D System (intraoral scanner with NIRI technology) and bitewing radiography (BWX). All evaluations will be carried out by 02 examiners. The examiners will be trained and calibrated to use the visual and radiographic criteria, and also to use the iTero 5D intraoral scanner, following the manufacturer's guidance.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes who seek dental treatment at the Dentistry Clinic of Universidade Metropolitana de Santos.
* Be between 04 and 10 years old;
* Good general health;
* Present at least two tooth surfaces that can be included in the study.

Exclusion Criteria:

* Dental surfaces with proximal restorations;
* Surfaces with evident proximal cavities (marginal crest break);
* Absence of adjacent tooth (absence of proximal contact).

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-01-20 (Estimated); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of primary caries lesions through visual inspection (ICDAS) | Baseline.
  For the visual inspection of caries, the International Caries Detection and Assessment System (ICDAS) evaluation system will be used. Complete ICDAS has seven categories, the first for healthy teeth (code 0) and the next two for limited enamel caries, white/brown stain (codes 1 and 2). The following two categories (codes 3 and 4) are considered to be caries that extend to the enamel without exposed dentin. And the two remaining categories (codes 5 and 6), are considered caries with exposed dentin.
Diagnosis of primary caries lesions through the iTero Element 5D scan | Baseline.
  For the diagnosis through scanning, the iTero 5D (Align Technology) equipment featuring NIRI Technology will be used. The Infrared Imaging Technology (NIRI) is a diagnostic tool that allows the detection of interproximal and occlusal caries in several stages, from the initial enamel caries to lesions in the amelo-dentin junction, without the use of ionizing radiation. Infrared is the region of the electromagnetic spectrum between 0.7 and 2.0 micrometers (µm). The iTero Element 5D imaging system uses wavelength light (= 850 nm) in an electromagnetic spectrum that, in interaction with the hard tooth tissue, provides additional data on its structure.
Diagnosis of primary caries lesions BWX Radiographic Assessment | Baseline.
  For this diagnosis, participants will be radiographed with a digital X-ray device (DIOX-602, Micro Imagem, Indaiatuba, Brazil) with a regulation of 60 kV and 2 mA and exposure time of 0.10s. The technique used will be the interproximal/bitewing (BWX), with the FIT T1 Digital Sensor (external dimensions: 36.7mm x 24.3mm/sensitive area dimensions: 30.0mm x 20.0mm - 600mm²) and the sockets will be standardized with use of Han-Shin radiographic positioners (Jon, São Paulo, Brazil).

REFERENCES:
- [Derived] Sobral APT, Goncalves MLL, D Annibale AS, Santos EM, Guedes CC, Gallo JMAS, Ferri EP, Moretti LAC, Motta LJ, Deana AM, Horliana ACRT, Kalil Bussadori S. Evaluation of different methods for the diagnosis of primary caries lesions: Study protocol for a randomized controlled clinical trial. PLoS One. 2022 Aug 24;17(8):e0273104. doi: 10.1371/journal.pone.0273104. eCollection 2022. PMID 36001544